CLINICAL TRIAL: NCT03628820
Title: Canine Assisted Therapy to Reduce Emergency Care Provider Stress
Acronym: CANINE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jeffrey Kline, Professor Emergency Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1804891471
Record Dates: First submitted 2018-07-18; First posted 2018-08-14 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Stress; Anxiety
Keywords: Stress; Anxiety; Cortisol; Therapy; Dog; Coloring; Mandala
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapy Dog (Experimental): This group is exposed to the therapy dog and handler. On a convenience sample of shifts, a dog will be available. Participants will not know when dogs will be present and will not be informed of whether or not they will see a dog on any given shift. The dog and handler will be kept out of site of other providers. Participants who agree to participate will be approached by study personnel between 3 and 7 hours into his or her shift and asked "would now be a good time to see a therapy dog?" If the physician answers yes, then the physician will be escorted to a separate private, quiet room away from the usual work area to interact with a therapy dog and handler. We will ask the physician to spend approximately 5 minutes with the therapy dog, but will not specify or mandate any time. Study personnel will record the time spent. Only the handler and dog will be present in the room.
  Interventions: Behavioral: Dog Therapy
- Mandala Coloring (Experimental): This group is not exposed to the therapy dog or handler. At 3-7 hours into the shift, study personnel will encourage providers to take a 5 min period of mindfulness, achieved by coloring mandalas. Participants will be escorted out of the work area to the same private, quiet room where the interaction occurs with the dog and handler in the therapy dog group. Participants will have their choice of one of three mandalas to color and will be provided a full palette of colored pencils. When the provider's time is up, study personnel will notify them of the five minute period. Study personnel will not be present in the room but will photograph the work when the participant is done with the session and record the image in REDcap. The original art work will be returned to the provider.
  Interventions: Behavioral: Coloring
- No Intervention (No Intervention): This group is not exposed to the therapy dog or handler.

INTERVENTIONS:
Behavioral: Dog Therapy — 5 minutes spent with therapy dog during shift
  Arms: Therapy Dog
Behavioral: Coloring — 5 minutes spend coloring mandalas during shift
  Arms: Mandala Coloring

SUMMARY:
The main study hypothesis is that emergency healthcare workers on shift who interact for 5 min with a therapy dog and handler will have lower perceived and manifested stress response compared with use of a time out that includes voluntary use of a coloring mandalas. The work will also address two exploratory hypotheses: The first is that salivary cortisol will correlate significantly with perceived stress and will increase from beginning to end of shift, and that exposure to a therapy dog will blunt this increase. The second exploratory hypothesis states that participants who interact with a therapy dog will display more empathic behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria require that participants work full time as either a nurse or physician in the Eskenazi emergency department and are willing to consent to participation.
* Participants will include residents, faculty and nurses who work in the emergency department

Exclusion Criteria:

* Exclusions include any reported prior fear or adverse reaction to dogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Cortisol change | 4 hours
  Time and location of shift and times of each measurement. T1: As soon as practicable at shift start: Baseline perceived stress scale and anxiety scale (shown below) and approximately 100 uL of saliva using a commercial kit (Salimetrics® 1-3002 (5PK 1-3002-5)). Saliva is collected > 10 min after any eating or drinking. T2: Repeat perceived stress scale, anxiety scale and saliva approximately 15-30 min after exposure to the dog and handler or the coloring.
  Scale 0 to 10
  0=balanced mood 2=slight fear and worry 4= mild fear and worry 6=moderate worry, physical agitation 8= strong agitation, pacing, can't sit still 10= out of control behavior, self-harm

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Indianapolis, Indiana, United States